CLINICAL TRIAL: NCT04428307
Title: Malaria Diagnostic Testing and Conditional Subsidies to Target ACTs in the Retail Sector: the TESTsmART Trial Aim 2
Brief Title: Malaria Diagnostic Testing and Conditional Subsidies to Target ACTs in the Retail Sector: TESTsmART Aim 2 - Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Moi University (Other); Clinton Health Access Initiative Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00104256; 5R01AI141444-02 (NIH)
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Malaria; Febrile Illness
Keywords: treatment seeking in the informal (retail) health sector; malaria diagnostic testing; rational drug use
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: three-arm parallel cluster randomized trial
Who Masked: Outcomes Assessor
Masking Description: Interviewers assessing outcomes and statisticians will be blinded to arm assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (control) (No Intervention): RDTs available at study-recommended price, providers trained on mobile reporting app
- Arm 2 (client-directed intervention) (Experimental): ACT subsidy to client conditional on positive RDT, RDTs available at study-recommended price
  Interventions: Other: Conditional artemisinin combination therapy subsidy
- Arm 3 (client-directed and provider-directed intervention) (Experimental): providers receive a small payment for each RDT that they perform and consumers with a positive test are eligible for a subsidy on a quality-assured ACT, RDTs are available at study recommended price
  Interventions: Other: Conditional artemisinin combination therapy subsidy; Other: Testing incentive

INTERVENTIONS:
Other: Conditional artemisinin combination therapy subsidy — An additional discount on WHO-approved quality assured ACTs will be offered to individuals with a positive RDT.
  Arms: Arm 2 (client-directed intervention); Arm 3 (client-directed and provider-directed intervention)
Other: Testing incentive — A small incentive will be paid to the provider each time they perform a malaria rapid diagnostic test.
  Arms: Arm 3 (client-directed and provider-directed intervention)

SUMMARY:
Highly subsidized first-line antimalarials (artemisinin combination therapy or ACT) are available over the counter in the private retail sector in most malaria-endemic countries. Overconsumption of ACTs purchased over the counter is rampant due to their low price, high perceived efficacy, and absence of diagnostic tools to guide drug use. The ultimate goal of the proposed work is to improve antimalarial stewardship in the retail sector, which is responsible for distributing the majority of antimalarials in sub-Saharan Africa. Through a combination of diagnosis and treatment subsidies and provider-directed incentives, this approach will align provider and customer incentives with appropriate case management and thereby improve health outcomes.

The main objective of this study (Aim 2) is to test two key interventions in a random sample of private medicine retail outlets in Kenya. This will be a cluster-randomized controlled trial where the cluster is a private retail outlet that stocks and sells WHO quality-assured ACTs. This three-arm study will test 1) a consumer-directed intervention in the form of a diagnosis-dependent ACT subsidy, 2) both a provider-directed incentive for testing and a client-directed intervention in combination against 3) a comparison arm. Outlets in all three arms will offer malaria diagnostic testing to customers who wish to purchase one. Information for the primary and secondary outcomes will be collected during exit interviews with eligible customers. The primary outcome will be the proportion of ACTs sold to customers with a positive diagnostic test. The main secondary outcome will be the proportion of suspected malaria cases presenting to the retail outlet that are tested. Other secondary outcomes include adherence to the RDT result amongst those tested (defined as taking a quality-assured ACT following a positive test and refraining from taking an ACT following a negative test) and appropriate case management for all suspected malaria cases (proportion tested and adhered among all suspected cases).

DETAILED DESCRIPTION:
RATIONALE:

The investigators hypothesize that decision-making in the retail sector is influenced primarily by price (or profit) supplemented by individual beliefs or preferences. Information from a diagnostic test, when available, plays only a minor role in the decision-making landscape. In response to this, the investigators propose to test a scalable, policy-relevant strategy that integrates testing and treatment subsidies and makes ACT subsidies available only to customers with a positive malaria test. Differential pricing based on the results of the diagnostic test will align consumer and provider incentives (price and profit) with testing and appropriate ACT use. This approach will also ensure that public subsidies are directed at confirmed malaria cases thereby enhancing the sustainability of such programs. By allocating subsidy dollars across both testing and conditional treatment (rather than universal, treatment-only subsidies), the investigators can reduce the cost of subsidizing malaria treatment and improve targeting of ACTs without compromising access.

OBJECTIVES:

This goal of the proposed work is to improve antimalarial stewardship in the retail sector, which has the largest market share of antimalarials in sub-Saharan Africa. In this study (Aim 2) the investigators will use a cluster randomized controlled trial to measure the impact of two innovative interventions - a provider-directed incentive for offering malaria rapid diagnostic tests to suspected malaria cases and a consumer-directed diagnosis dependent ACT subsidy (conditional ACT subsidy). The unit of randomization will be the private medicine outlet (cluster).

STUDY DESIGN:

The study will be a cluster-randomized controlled trial with three arms. The original study design was for a four-arm trial (an additional arm that would have tested the provider-directed incentive alone), however preliminary data from the study area indicated that the study may not be powered to measure the effect of a four arm study. No participants were enrolled prior to finalization of the study design, and all clusters will be randomized to one of the three remaining study arms only (1) control, 2) client-directed intervention, and 3) combined client- and provider-directed intervention). See Section 4.4 Statistical Design and Power for complete detail.

STUDY POPULATION:

The study will be conducted in Kenya, a country with high malaria burden. Kenya has the programmatic goal of universal access to prompt parasitological confirmation before treatment and have endorsed the use of malaria RDTs in the public health sector at all levels of care. However, very high rates of treatment in the retail sector undermine the explicit policy that all malaria cases should be confirmed by parasitological diagnosis. In Kenya, retail outlets currently do not conduct RDTs and emphasis has been placed on implementing community case management for malaria through public-sector community health workers (including conducting RDTs).

The specific study site will be western Kenya (Bungoma County and Trans Nzoia county).

STUDY PROCEDURES:

A complete sampling frame of eligible retail outlets will be made for the site. Outlets will be eligible if they regularly carry quality-assured, subsidized ACTs. Attendants who dispense medicines at each outlet will be trained to correctly and safely perform RDTs. They will receive an initial small start-up stock of RDTs and will be given contact information for RDT wholesalers who can provide replenishment stocks on demand. In addition, all attendants will be trained to use a mobile reporting app that captures basic information about suspected malaria cases. This app will not be used to assess outcomes, but will be an important monitoring tool and serve as the conduit for all payments according to the arm assignment.

Following training, shops will be randomized to one of the three arms:

* Arm 1 (control): RDTs available at study-recommended price, providers trained on mobile app
* Arm 2 (client-directed intervention): ACT subsidy to client conditional on positive RDT, RDTs available at study-recommended price
* Arm 3 (client-directed and provider-directed intervention): providers are reimbursed for each RDT and consumers with a positive test are eligible for a subsidy on a quality-assured ACT. RDTs are available at study recommended price.

Customers who come to a participating outlet in any arm with fever or suspected malaria are eligible for an RDT at the study-recommended price and, in arms 2 and 3, a conditional ACT subsidy when the RDT is positive. Attendants will be trained to recognize danger signs and refer those individuals to a health facility for immediate care. Customers purchasing medicine on someone's behalf or those who have already had a malaria test will not be eligible for RDT testing or conditional subsidies.

Study outcome measures will be collected by interviewing a random sample of customers leaving participating shops (exit interviews). A team of field interviewers will be trained in each site and will be assigned to participating outlets on random days in a month. Both the day of the month and the interviewer assigned to the specific outlet will be randomized in order to balance data collection across interviewers and arms and to minimize the observer effect. Each outlet will be visited thrice in a month and the interviewer will enroll eligible participants in succession until they have completed 3-4 interviews. Ten customers per month per outlet are needed to reach a sample size of 170 interviews per outlet in 15 months of data collection. Exit interviews will capture information about customer demographics, symptoms of their current illness, whether they had a malaria diagnostic test at the outlet or elsewhere, how much they paid for the test, the results of the test, and the drug(s) they purchased. Customers will be eligible to participate in the exit interview if s/he was seeking drugs for him/herself or their minor child older than one year of age and the child is physically present, s/he had a febrile illness or suspected malaria, and s/he agrees to be interviewed.

Study monitoring will be continuous throughout the study period using the mobile app. Study staff will regularly review reporting data captured by the mobile app. In particular, pictures of RDTs will be reviewed alongside results reported by outlet attendants to ensure correct use and interpretation of the RDTs. In addition, exit interviews will be summarized monthly by outlet and compared to the data submitted via the app. This monitoring step will allow us to identify major discrepancies between actions reported by the shop and those reported by the customers such as testing rates, RDT positivity rates, dispensing of qualified ACTs and prices charged for RDTs and ACTs.

SAMPLE SIZE AND POWER:

The investigators calculated power based on a cluster randomized two-sample two-tailed t-test for the comparison of two proportions. The investigators calculated power for differences in the primary outcome for each of the two comparisons of interest noted above. With a sample of 170 exit interviews per outlet (40 outlets in Kenya), the investigators will have >90% power to detect a minimum difference between Arms 1 (control) and 3 (combined interventions) in the primary outcome of 16 percentage points. The investigators will also have >80% power to detect a minimum difference of 11 percentage points for the main secondary comparison of interest (testing uptake).

The sample size estimates correspond to a total of 6800 exit interviews with clients in Kenya. Since not everyone interviewed will have purchased an ACT, estimates account for the fact that only a subset will enter into the analysis for the primary outcome. The investigators will have a team of 8 data collectors and each data collector will conduct approximately 50-60 interviews per month. Exit interviews should take 15 months to complete.

See Section 4.4 Statistical Design and Power for comprehensive description of sample size, power and statistical analysis.

SUBJECT CONFIDENTIALITY:

Customers leaving the shop will be approached by the field interviewer to ask if they are interested in participating in a short interview. If they agree, then they will be taken to a private area and the study will be explained to them. Once they provide consent, the interviewer will record the details of their illness and treatment at the outlet. No participant identifiers will be recorded in the electronic data collection form. This limits the possibility of identifying the source of any health information (See Protection of Human Subjects Section 3.3).

ELIGIBILITY:
All clients attending a participating outlet on the day selected for exit interviews will be eligible to be screened for inclusion into the interview sample.

Inclusion Criteria:

* Participants with fever, or history of fever in the last 48 hours, or suspects they may have malaria
* Individual with malaria-like illness must be present at recruitment
* Older than one year of age

Exclusion Criteria:

* Any individual with signs of severe illness requiring immediate referral
* Individuals who have taken an antimalarial in the last seven days, including for the current illness
* Patients <18 years without a parent or legal guardian present

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5696 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy P O'Meara, PhD, Principal Investigator — Duke University
Locations (1):
- Moi University, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Visser T, Laktabai J, Kimachas E, Kipkoech J, Menya D, Arthur D, Zhou Y, Chepkwony T, Abel L, Robie E, Amunga M, Ambani G, Uhomoibhi P, Ogbulafor N, Oshinowo B, Ogunsola O, Woldeghebriel M, Garber E, Olaleye T, Eze N, Nwidae L, Mudabai P, Gallis JA, Fashanu C, Saran I, Woolsey A, Turner EL, Prudhomme O'Meara W. A cluster-randomized trial of client and provider directed financial interventions to align incentives with appropriate case management in private medicine retailers: results of the TESTsmART Trial in Lagos, Nigeria. medRxiv [Preprint]. 2024 Jan 31:2024.01.30.24302026. doi: 10.1101/2024.01.30.24302026. PMID 38352390
- [Derived] Laktabai J, Kimachas E, Kipkoech J, Menya D, Arthur D, Zhou Y, Chepkwony T, Abel L, Robie E, Amunga M, Ambani G, Woldeghebriel M, Garber E, Eze N, Mudabai P, Gallis JA, Fashanu C, Saran I, Woolsey A, Visser T, Turner EL, Prudhomme O'Meara W. A cluster-randomized trial of client and provider-directed financial interventions to align incentives with appropriate case management in retail medicine outlets: Results of the TESTsmART Trial in western Kenya. PLOS Glob Public Health. 2024 Feb 7;4(2):e0002451. doi: 10.1371/journal.pgph.0002451. eCollection 2024. PMID 38324584
- [Derived] Woolsey AM, Simmons RA, Woldeghebriel M, Zhou Y, Ogunsola O, Laing S, Olaleye T, Kipkoech J, Rojas BM, Saran I, Odhiambo M, Malinga J, Ambani G, Kimachas E, Fashanu C, Wiwa O, Menya D, Laktabai J, Visser T, Turner EL, O'Meara WP. Incentivizing appropriate malaria case management in the private sector: a study protocol for two linked cluster randomized controlled trials to evaluate provider- and client-focused interventions in western Kenya and Lagos, Nigeria. Implement Sci. 2021 Jan 20;16(1):14. doi: 10.1186/s13012-020-01077-w. PMID 33472650

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between Jan 2021 and August 2022, with customers leaving participating outlets screened for study eligibility by trained exit interviewers.
Pre-assignment Details: Participating shops were randomly assigned to each arm of the study, with the exception of 2 pairs of shops that were within visual distance of each other and therefore assigned to the same study arm.
Units Other Than Participants: Retail medicine outlets
Period: Overall Study
Arm/Group | Arm 1 (Control) | Arm 2 (Client-directed Intervention) | Arm 3 (Client-directed and Provider-directed Intervention)
Started | 1692; 13 Retail medicine outlets | 1789; 13 Retail medicine outlets | 2215; 13 Retail medicine outlets
Completed | 1692; 13 Retail medicine outlets | 1789; 13 Retail medicine outlets | 2214; 13 Retail medicine outlets
Not Completed | 0; 0 Retail medicine outlets | 0; 0 Retail medicine outlets | 1; 0 Retail medicine outlets

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Control) | Arm 2 (Client-directed Intervention) | Arm 3 (Client-directed and Provider-directed Intervention) | Total
Number analyzed (Participants) | 1692 | 1789 | 2214 | 5695
Age, Customized [Count of Participants; unit: Participants]
  Age in years: 18-25 | 264 | 263 | 314 | 841
  Age in years: 26-39 | 672 | 719 | 922 | 2313
  Age in years: 40-59 | 579 | 622 | 766 | 1967
  Age in years: 60-79 | 160 | 167 | 196 | 523
  Age in years: 80+ | 13 | 15 | 10 | 38
  Age in years: Unknown | 4 | 3 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender missing for 1 participant in Arm 2 and 4 participants in Arm 3.
  Participants
    number analyzed (Participants) | 1692 | 1788 | 2210 | 5690
    Female | 939 | 968 | 1262 | 3169
    Male | 753 | 820 | 948 | 2521
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1692 | 1789 | 2214 | 5695
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1692 | 1789 | 2214 | 5695
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Kenya | 1692 | 1789 | 2214 | 5695

OUTCOME MEASURES:

1. Primary Outcome: ACT (Artemisinin Combination Therapy) Consumption by True Malaria Cases
Description: Number of participants who purchased ACTs and were malaria test-positive. Malaria test-positivity was based on mRDT testing testing at the outlet or documented testing brought to the facility.
Time Frame: Day of enrollment
Population: Participants who purchased ACTs.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Control) | Arm 2 (Client-directed Intervention) | Arm 3 (Client-directed and Provider-directed Intervention)
Number analyzed (Participants) | 1039 | 1004 | 1293
Participants | 313 | 250 | 339
Statistical Analysis 1: Comparison: Arm 1 (Control) vs Arm 3 (Client-directed and Provider-directed Intervention); Test type: Superiority; Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.61 to 2.02]
Statistical Analysis 2: Comparison: Arm 2 (Client-directed Intervention) vs Arm 3 (Client-directed and Provider-directed Intervention); Test type: Superiority; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.49 to 1.71]

2. Secondary Outcome: Use of Malaria Rapid Diagnostic Test
Description: Number of participants with suspected malaria cases presenting to the retail outlet that are tested.
Time Frame: Day of enrollment
Population: Only participants who were suspected of having malaria were included in this analysis. This included anyone who tested for malaria or purchased antimalarials without a test.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Control) | Arm 2 (Client-directed Intervention) | Arm 3 (Client-directed and Provider-directed Intervention)
Number analyzed (Participants) | 1541 | 1576 | 1878
Participants | 819 | 804 | 813
Statistical Analysis 1: Comparison: Arm 1 (Control) vs Arm 3 (Client-directed and Provider-directed Intervention); Test type: Superiority; Risk Ratio (RR) = 1.22, 95% CI 2-sided [0.83 to 1.80]
Statistical Analysis 2: Comparison: Arm 2 (Client-directed Intervention) vs Arm 3 (Client-directed and Provider-directed Intervention); Test type: Superiority; Risk Ratio (RR) = 1.15, 95% CI 2-sided [0.81 to 1.62]

3. Secondary Outcome: Adherence to the RDT (Rapid Diagnostic Test) Result Among All Those Tested in the Shop
Description: The number of tested participants who are adherent where adherence to the test result is defined as taking a quality-assured ACT if the RDT is positive or taking another drug (or no drug) if the test is negative.
Time Frame: Day of enrollment
Population: Participants who tested at the outlet.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Control) | Arm 2 (Client-directed Intervention) | Arm 3 (Client-directed and Provider-directed Intervention)
Number analyzed (Participants) | 819 | 804 | 813
Participants | 558 | 595 | 591
Statistical Analysis 1: Comparison: Arm 1 (Control) vs Arm 3 (Client-directed and Provider-directed Intervention); Test type: Superiority; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.80 to 1.09]
Statistical Analysis 2: Comparison: Arm 2 (Client-directed Intervention) vs Arm 3 (Client-directed and Provider-directed Intervention); Test type: Superiority; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.85 to 1.16]

4. Secondary Outcome: Appropriate Case Management
Description: Number of all participants with suspected malaria cases that are managed appropriately (tested for malaria, and use ACT following a positive test and do not purchase an ACT after a negative test)
Time Frame: Day of enrollment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Control) | Arm 2 (Client-directed Intervention) | Arm 3 (Client-directed and Provider-directed Intervention)
Number analyzed (Participants) | 1541 | 1576 | 1878
Participants | 558 | 595 | 591
Statistical Analysis 1: Comparison: Arm 1 (Control) vs Arm 3 (Client-directed and Provider-directed Intervention); Test type: Superiority; Risk Ratio (RR) = 1.14, 95% CI 2-sided [0.75 to 1.73]
Statistical Analysis 2: Comparison: Arm 2 (Client-directed Intervention) vs Arm 3 (Client-directed and Provider-directed Intervention); Test type: Superiority; Risk Ratio (RR) = 1.15, 95% CI 2-sided [0.77 to 1.74]

5. Secondary Outcome: ACT (Artemisinin Combination Therapy) Use Among Untested Clients
Description: Number of participants who are not tested for malaria and purchased an ACT, among those who did not test in the shop, do not have documentation of a test, and purchased any antimalarial at the shop.
Time Frame: Day of enrollment
Population: Only participants who purchased any antimalarial without documented test results available were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Control) | Arm 2 (Client-directed Intervention) | Arm 3 (Client-directed and Provider-directed Intervention)
Number analyzed (Participants) | 676 | 746 | 798
Participants | 523 | 542 | 601
Statistical Analysis 1: Comparison: Arm 1 (Control) vs Arm 3 (Client-directed and Provider-directed Intervention); Test type: Superiority; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.95 to 1.11]
Statistical Analysis 2: Comparison: Arm 2 (Client-directed Intervention) vs Arm 3 (Client-directed and Provider-directed Intervention); Test type: Superiority; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.89 to 1.04]

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected.
Description: Adverse event data were not collected.
Arm/Group | Arm 1 (Control) | Arm 2 (Client-directed Intervention) | Arm 3 (Client-directed and Provider-directed Intervention)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT04428307/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT04428307/ICF_000.pdf